CLINICAL TRIAL: NCT04500223
Title: The Effect of Neck Stabilization Exercise Plus Cardiopulmonary Rehabilitation on Pulmonary Function of SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taoyuan General Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TYGH108045
Record Dates: First submitted 2020-05-07; First posted 2020-08-05 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Spinal Cord Injury
Keywords: Cervical exercise; Cardiopulmonary rehabilitation; Pulmonary function
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical Cranioflexion exercise plus cardiopulmonary exercise (Experimental): subjects who received Cervical Cranioflexion exercise plus cardiopulmonary exercise
  Interventions: Other: Cervical Cranioflexion exercise plus cardiopulmonary exercise
- Cervical stretch exercise plus cardiopulmonary rehabilitation (Active Comparator): subjects who received Cervical stretch exercise plus cardiopulmonary rehabilitation
  Interventions: Other: Cervical stretch exercise plus cardiopulmonary rehabilitation

INTERVENTIONS:
Other: Cervical Cranioflexion exercise plus cardiopulmonary exercise — Intervention:Cervical Cranioflexion exercise plus cardiopulmonary exercise
  Arms: Cervical Cranioflexion exercise plus cardiopulmonary exercise
Other: Cervical stretch exercise plus cardiopulmonary rehabilitation — control:Cervical stretch exercise plus cardiopulmonary rehabilitation
  Arms: Cervical stretch exercise plus cardiopulmonary rehabilitation

SUMMARY:
Cervicocranial flexion exercise (CCFE) and superficial neck flexor endurance training have been widely implemented in clinical practice for curing chronic neck pain. By means of CCFE, the muscle balance between deep neck flexor and superficial flexor would be optimal during neck movement. In other words, the superficial neck flexor( scalenes, SCM, and trapezius) would not overactive and the fatigue threshold might increase. Superficial neck flexor endurance training is proved to be efficient in reducing superficial cervical flexor muscle fatigue as well as increasing cervical flexion strength.

Reasonably, Cervicocranial flexion exercise (CCFE) and superficial neck flexor endurance training are also beneficial to pulmonary function due to training the respiratory accessory muscle (scalens and SCM). Hence this article hypothesizes that Cervicocranial flexion exercise (CCFE) and superficial neck flexor endurance training combined with common pulmonary rehabilitation will manifest better outcomes (pulmonary function, dyspnea situation, pain and stiffness level of neck) than pulmonary rehabilitation only.

DETAILED DESCRIPTION:
2.1 subject 20 patients were recruited in this article during 2020/03 to 2021/02. The inclusion criteria were 1.) SCI onset in a year; 2.) motor level above T12 and American Spinal Injury Association Impairment Scale (AIS) grade A, B, C, or D; 3.) age from 20~70; 4.) FEV1< 80% prediction value. The exclusion criteria were 1.) ventilation dependence 2.) Tracheostomy 3.) Psychiatric condition 4.) Progressive diseases 5.) infection 6.) cancer 7.)unable to speak Chinese or English. Patient who met the criteria would were asked to provide written informed consent. The IRB were approved by Tao Yuan General Hospital, Ministry of Health and Welfare, IRB committee.(TYGH108045 ) 2.2 procedure The subjects included in this study were randomized assigned to experimental group and control group. The randomization orders were decided by computer, and all the contents were concealed into a dark color envelop. Before first treatment, the envelops were opened to determine which treatment protocol were adopted. The treatment of experimental group was consist of Cervicocranial flexion exercise (CCFE) and neck flexor endurance training plus normal cardiopulmonary rehabilitation. The treatment of control group was composed of general neck stretch exercise plus cardiopulmonary rehabilitation. Subsequently, initial measurement was conducted including lung capacity test, dyspnea situation, pain and stiffness of neck. Moreover, lung function such as FVC and FEV1, dyspnea situation, pain and stiffness of neck were also recorded one time in a week as a short-term outcome. Then, the treatment protocols were both executed for 30 minutes, ten times in a month. After completing the treatment process, the final measurement were conducted as the initial treatment. All the outcome were collected and analyzed by statistically method.

2.3 Outcome measurement Lung capacity was evaluated by in lung function examination center of Taoyaun general hospital. The parameters revealed by this test. Before the examination, bronchodilator should not be used to avoid interfering the outcome of examination. In addition, portable lung capacity device(ezOxygen, Taipei, Taiwan) were adopted to record lung function parameters such as FVC and FEV1. First, subjects were instructed to hold deep breath and let his mouth firmly contact to the mouthpiece. Second, subjects were asked to exhale the air into the mouth and the process was repeated three times, between each sessions, subjects were allowed to rest at least thirty seconds. Three tests were recorded and the mean value was calculated. The dyspnea situation was evaluated by the questionnaire Baseline Dyspnea Index (BDI) and Transition Dyspnea Index (TDI). The BDI measured the severity of dyspnea at the baseline and the TDI measured the change from baseline. Both questionnaires are composed of three parts: functional impairment, magnitude of task, and magnitude of effort required to evoke dyspnea. Each part in BDI is scored from 0(very severe) to 4(no impairment) and total score from 0~12( the lower the score, the worse the severity of dyspnea) is also recorded. Each component in TDI is rated by seven grades ranging from -3 (major deterioration) to +3 (major improvement). Total score ranged from - 9 to + 9. The lower the score is, the more deterioration of the severity of dyspnea revealed. The minimal clinical important difference(MCID) of TDI is ≥1 unit[31]. The number rating scale NRS is used to define the level of neck pain and stiffness. The MCID of neck pain VAS is 1.5.

2.4 Treatment Experimental group is consist of CCFE and neck flexor endurance training plus normal cardiopulmonary rehabilitation. Subjects were instructed to perform chin in without excessive SCM contraction. CCFE was conducted in supine position. Subjects were asked to maintain chin for 10 seconds each repetition, ten repetitions for a set, 3 sets in a treatment session[30]. The physiotherapist with abundant experience related to CCFE supervised all the treatment process to confirm the quality of execution. If no symptoms revealed, the neck endurance exercise would involve into the treatment sessions. Neck endurance exercise was also conducted in supine position. Subjects were taught to lift their head with a neutral upper cervical spine first. Then, they gradually move the head and neck through as full range as possible without induce discomfort or neck related symptom. This exercise was performed 12~15 repetition depends on patient's condition[33]. If the subjects were unable to achieve the training level, subject's bed were inclined up from horizontal. Hence, the demand of lifting neck and head declined and subjects could perform aimed repetitions. The cardiopulmonary rehabilitation protocol was based on Wu, Y.-T. et al[9], and it was divide into three stages. In first stage, subjects lied in supine position, and they were instructed to do diaphragm breath, pursed-lip breath, lateral coastal breath, cough training, and rib mobilization. The dosage and type of therapy was decided depending on subjects situation everyday. The total cardiopulmonary training was controlled in 20 minutes. In second stage, the incentive spirometer (picture A) was integrated into the therapy. Subjects were asked to inhale the air slowly with eye contact at the chamber of the spirometer for controlling the air flow velocity. Subject were also asked to inhale as many volumes as possible. Back support was inclined to hold subject in semi-sitting position. 15 repetitions was given to subjects and subjects received 20 second rest between each repetition. In addition, some upper extremities training combined with breath exercise were also involved in after incentive spirometer training. 15 repetitions, 3 sets was given to subjects. In stage 3, the upper extremities exercise were combined with spirometer training. 15 repetitions, 3 sets was given to subjects. The experienced physiotherapist decided the stages depends on patient's capability, that is, the stages were not the same for every subject. The control group were composed of neck stretch exercise plus cardiopulmonary rehabilitation. The neck stretch exercises were executed by physiotherapist before cardiopulmonary training. Neck flexion, neck extension, neck right rotation, neck left rotation, neck right side-bending, and neck left side-bending were applied to subjects 5 times for each direction, and neck maintained at end position for 30 seconds each time.

2.5 Statistical analysis The primary variable of the study were vital capacity, respiratory complication ,and dyspnea. The secondary variable of the study were FEV1, pain and stiffness of neck. Descriptive statistics for the categorical variable were documented as frequency counts and percentages. The continuous variables were reported as mean + SD, if they were normal distribution, or they were recorded as median and range.

The Wilcox signed test was adopted to analyze the treatment before and after the treatment sessions (time effect). The Mann-Whitney U was applied for the difference before and after treatment between two groups (group effect), and the baseline of two groups was also analyzed by this method. The significant level was set as p value< 0.05. All the statistical data analysis were performed by SPSS version 22.

ELIGIBILITY:
Inclusion Criteria:

* SCI onset in a year.
* Motor level above T12 and American Spinal Injury Association Impairment Scale (AIS) grade A, B, C, or D.
* Age from 20~70.
* FEV1< 80% prediction value.

Exclusion Criteria:

* Ventilation dependent
* Tracheostomy
* Psychiatric condition
* Progressive diseases
* infection
* Cancer
* Unable to speak Chinese or English.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
FVC change | initial points, first week, second week, final points.(total 3 week)
  liter
FEV1/FVC change | initial points, first week, second week, final points.(total 3 week)
  percentage
Baseline Dyspnea Index (BDI) and Transition Dyspnea Index (TDI) score change | initial points, first week, second week, final points.(total 3 week)
  points

CONTACTS AND LOCATIONS:
Locations (1):
- Taoyaun General Hospital, Ministry of Wealth and Health, Taoyuan District, Taoyuan Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burns AS, Marino RJ, Flanders AE, Flett H. Clinical diagnosis and prognosis following spinal cord injury. Handb Clin Neurol. 2012;109:47-62. doi: 10.1016/B978-0-444-52137-8.00003-6. PMID 23098705
- [Background] Brown R, DiMarco AF, Hoit JD, Garshick E. Respiratory dysfunction and management in spinal cord injury. Respir Care. 2006 Aug;51(8):853-68;discussion 869-70. PMID 16867197
- [Background] Mueller G, de Groot S, van der Woude L, Hopman MT. Time-courses of lung function and respiratory muscle pressure generating capacity after spinal cord injury: a prospective cohort study. J Rehabil Med. 2008 Apr;40(4):269-76. doi: 10.2340/16501977-0162. PMID 18382822
- [Background] Fishburn MJ, Marino RJ, Ditunno JF Jr. Atelectasis and pneumonia in acute spinal cord injury. Arch Phys Med Rehabil. 1990 Mar;71(3):197-200. PMID 2317137
- [Background] Reines HD, Harris RC. Pulmonary complications of acute spinal cord injuries. Neurosurgery. 1987 Aug;21(2):193-6. doi: 10.1227/00006123-198708000-00010. PMID 3658131
- [Background] van den Berg ME, Castellote JM, de Pedro-Cuesta J, Mahillo-Fernandez I. Survival after spinal cord injury: a systematic review. J Neurotrauma. 2010 Aug;27(8):1517-28. doi: 10.1089/neu.2009.1138. PMID 20486810
- [Background] Schilero GJ, Spungen AM, Bauman WA, Radulovic M, Lesser M. Pulmonary function and spinal cord injury. Respir Physiol Neurobiol. 2009 May 15;166(3):129-41. doi: 10.1016/j.resp.2009.04.002. Epub 2009 Apr 9. PMID 19442929
- [Background] Fawcett JW, Curt A, Steeves JD, Coleman WP, Tuszynski MH, Lammertse D, Bartlett PF, Blight AR, Dietz V, Ditunno J, Dobkin BH, Havton LA, Ellaway PH, Fehlings MG, Privat A, Grossman R, Guest JD, Kleitman N, Nakamura M, Gaviria M, Short D. Guidelines for the conduct of clinical trials for spinal cord injury as developed by the ICCP panel: spontaneous recovery after spinal cord injury and statistical power needed for therapeutic clinical trials. Spinal Cord. 2007 Mar;45(3):190-205. doi: 10.1038/sj.sc.3102007. Epub 2006 Dec 19. PMID 17179973
- [Background] Wu, Y.-T., 脊髓損傷病人的呼吸功能復健, in Cardiopulmonary Physical Therapy-Basic to practice-second edition. 2012: Taiwan. p. 417~432
- [Background] Hopman MT, van der Woude LH, Dallmeijer AJ, Snoek G, Folgering HT. Respiratory muscle strength and endurance in individuals with tetraplegia. Spinal Cord. 1997 Feb;35(2):104-8. doi: 10.1038/sj.sc.3100353. PMID 9044518
- [Background] Mateus SR, Beraldo PS, Horan TA. Maximal static mouth respiratory pressure in spinal cord injured patients: correlation with motor level. Spinal Cord. 2007 Aug;45(8):569-75. doi: 10.1038/sj.sc.3101998. Epub 2006 Nov 28. PMID 17130889
- [Background] Liaw MY, Lin MC, Cheng PT, Wong MK, Tang FT. Resistive inspiratory muscle training: its effectiveness in patients with acute complete cervical cord injury. Arch Phys Med Rehabil. 2000 Jun;81(6):752-6. doi: 10.1016/s0003-9993(00)90106-0. PMID 10857519
- [Background] Berlowitz DJ, Tamplin J. Respiratory muscle training for cervical spinal cord injury. Cochrane Database Syst Rev. 2013 Jul 23;2013(7):CD008507. doi: 10.1002/14651858.CD008507.pub2. PMID 23881660
- [Background] Hart JE, Goldstein R, Walia P, Teylan M, Lazzari A, Tun CG, Garshick E. FEV1 and FVC and systemic inflammation in a spinal cord injury cohort. BMC Pulm Med. 2017 Aug 15;17(1):113. doi: 10.1186/s12890-017-0459-6. PMID 28810847
- [Background] Garshick E, Mulroy S, Graves DE, Greenwald K, Horton JA, Morse LR. Active Lifestyle Is Associated With Reduced Dyspnea and Greater Life Satisfaction in Spinal Cord Injury. Arch Phys Med Rehabil. 2016 Oct;97(10):1721-7. doi: 10.1016/j.apmr.2016.02.010. Epub 2016 Mar 4. PMID 26951870
- [Background] Sinderby C, Ingvarsson P, Sullivan L, Wickstrom I, Lindstrom L. Electromyographic registration of diaphragmatic fatigue during sustained trunk flexion in cervical cord injured patients. Paraplegia. 1992 Sep;30(9):669-77. doi: 10.1038/sc.1992.131. PMID 1408345
- [Background] Taylor BJ, West CR, Romer LM. No effect of arm-crank exercise on diaphragmatic fatigue or ventilatory constraint in Paralympic athletes with cervical spinal cord injury. J Appl Physiol (1985). 2010 Aug;109(2):358-66. doi: 10.1152/japplphysiol.00227.2010. Epub 2010 May 20. PMID 20489038
- [Background] Van Houtte S, Vanlandewijck Y, Gosselink R. Respiratory muscle training in persons with spinal cord injury: a systematic review. Respir Med. 2006 Nov;100(11):1886-95. doi: 10.1016/j.rmed.2006.02.029. Epub 2006 Apr 12. PMID 16626951
- [Background] Shin JC, Han EY, Cho KH, Im SH. Improvement in Pulmonary Function with Short-term Rehabilitation Treatment in Spinal Cord Injury Patients. Sci Rep. 2019 Nov 19;9(1):17091. doi: 10.1038/s41598-019-52526-6. PMID 31745108
- [Background] Lin KH, Lai YL, Wu HD, Wang TQ, Wang YH. Cough threshold in people with spinal cord injuries. Phys Ther. 1999 Nov;79(11):1026-31. PMID 10534795
- [Background] Reid WD, Brown JA, Konnyu KJ, Rurak JM, Sakakibara BM. Physiotherapy secretion removal techniques in people with spinal cord injury: a systematic review. J Spinal Cord Med. 2010;33(4):353-70. doi: 10.1080/10790268.2010.11689714. PMID 21061895
- [Background] Viroslav J, Rosenblatt R, Tomazevic SM. Respiratory management, survival, and quality of life for high-level traumatic tetraplegics. Respir Care Clin N Am. 1996 Jun;2(2):313-22. PMID 9390885
- [Background] James WS 3rd, Minh VD, Minteer MA, Moser KM. Cervical accessory respiratory muscle function in a patient with a high cervical cord lesion. Chest. 1977 Jan;71(1):59-64. doi: 10.1378/chest.71.1.59. PMID 830501
- [Background] Terson de Paleville D, Lorenz D. Compensatory muscle activation during forced respiratory tasks in individuals with chronic spinal cord injury. Respir Physiol Neurobiol. 2015 Oct;217:54-62. doi: 10.1016/j.resp.2015.07.001. Epub 2015 Jul 11. PMID 26169572
- [Background] Falla D, Jull G, Hodges P, Vicenzino B. An endurance-strength training regime is effective in reducing myoelectric manifestations of cervical flexor muscle fatigue in females with chronic neck pain. Clin Neurophysiol. 2006 Apr;117(4):828-37. doi: 10.1016/j.clinph.2005.12.025. Epub 2006 Feb 21. PMID 16490395
- [Background] Falla D, Jull G, Rainoldi A, Merletti R. Neck flexor muscle fatigue is side specific in patients with unilateral neck pain. Eur J Pain. 2004 Feb;8(1):71-7. doi: 10.1016/S1090-3801(03)00075-2. PMID 14690677
- [Background] Borisut S, Vongsirinavarat M, Vachalathiti R, Sakulsriprasert P. Effects of strength and endurance training of superficial and deep neck muscles on muscle activities and pain levels of females with chronic neck pain. J Phys Ther Sci. 2013 Sep;25(9):1157-62. doi: 10.1589/jpts.25.1157. Epub 2013 Oct 20. PMID 24259936
- [Background] Ghaderi F, Jafarabadi MA, Javanshir K. The clinical and EMG assessment of the effects of stabilization exercise on nonspecific chronic neck pain: A randomized controlled trial. J Back Musculoskelet Rehabil. 2017;30(2):211-219. doi: 10.3233/BMR-160735. PMID 27472855
- [Background] Jull G, Falla D. Does increased superficial neck flexor activity in the craniocervical flexion test reflect reduced deep flexor activity in people with neck pain? Man Ther. 2016 Sep;25:43-7. doi: 10.1016/j.math.2016.05.336. Epub 2016 Jun 4. PMID 27422596
- [Background] Jull GA, Falla D, Vicenzino B, Hodges PW. The effect of therapeutic exercise on activation of the deep cervical flexor muscles in people with chronic neck pain. Man Ther. 2009 Dec;14(6):696-701. doi: 10.1016/j.math.2009.05.004. Epub 2009 Jul 25. PMID 19632880
- [Background] Witek TJ Jr, Mahler DA. Minimal important difference of the transition dyspnoea index in a multinational clinical trial. Eur Respir J. 2003 Feb;21(2):267-72. doi: 10.1183/09031936.03.00068503a. PMID 12608440
- [Background] Katch, W.D.M.F.I.K.V.L., Exercise physiology. 1996
- [Background] Kovacs FM, Abraira V, Royuela A, Corcoll J, Alegre L, Tomas M, Mir MA, Cano A, Muriel A, Zamora J, Del Real MT, Gestoso M, Mufraggi N; Spanish Back Pain Research Network. Minimum detectable and minimal clinically important changes for pain in patients with nonspecific neck pain. BMC Musculoskelet Disord. 2008 Apr 10;9:43. doi: 10.1186/1471-2474-9-43. PMID 18402665
- [Derived] Tsai CS, Li HT, Yang WL, Jhan YT. The effect of craniocervical flexion and neck endurance exercises plus pulmonary rehabilitation on pulmonary function in spinal cord injury: a pilot single-blinded randomised controlled trial. Spinal Cord Ser Cases. 2024 Apr 23;10(1):27. doi: 10.1038/s41394-024-00637-2. PMID 38654004